CLINICAL TRIAL: NCT02173535
Title: Quantitative Study of New Limbal Ring Prototypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR-5590
Record Dates: First submitted 2014-05-20; First posted 2014-06-25 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Cosmetic Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- etafilcon test contact lens Variant AP (Experimental)
  Interventions: Device: etafilcon test contact lens Variant AP; Device: etafilcon test contact lens Variant JG; Device: etafilcon test contact lens Variant CS; Device: etafilcon test contact lens Variant VC; Device: etafilcon test contact lens Variant LA
- etafilcon test contact lens Variant JG (Experimental)
  Interventions: Device: etafilcon test contact lens Variant AP; Device: etafilcon test contact lens Variant JG; Device: etafilcon test contact lens Variant CS; Device: etafilcon test contact lens Variant VC; Device: etafilcon test contact lens Variant LA
- etafilcon test contact lens Variant CS (Experimental)
  Interventions: Device: etafilcon test contact lens Variant AP; Device: etafilcon test contact lens Variant JG; Device: etafilcon test contact lens Variant CS; Device: etafilcon test contact lens Variant VC; Device: etafilcon test contact lens Variant LA
- etafilcon test contact lens Variant VC (Experimental)
  Interventions: Device: etafilcon test contact lens Variant AP; Device: etafilcon test contact lens Variant JG; Device: etafilcon test contact lens Variant CS; Device: etafilcon test contact lens Variant VC; Device: etafilcon test contact lens Variant LA
- etafilcon test contact lens Variant LA (Experimental)
  Interventions: Device: etafilcon test contact lens Variant AP; Device: etafilcon test contact lens Variant JG; Device: etafilcon test contact lens Variant CS; Device: etafilcon test contact lens Variant VC; Device: etafilcon test contact lens Variant LA

INTERVENTIONS:
Device: etafilcon test contact lens Variant AP — Subject will complete a questionnaire regarding cosmetic effect of the lens post insertion, then remove the lens.
Device: etafilcon test contact lens Variant JG — Subject will complete a questionnaire regarding cosmetic effect of the lens post insertion, then remove the lens.
Device: etafilcon test contact lens Variant CS — Subject will complete a questionnaire regarding cosmetic effect of the lens post insertion, then remove the lens.
Device: etafilcon test contact lens Variant VC — Subject will complete a questionnaire regarding cosmetic effect of the lens post insertion, then remove the lens.
Device: etafilcon test contact lens Variant LA — Subject will complete a questionnaire regarding cosmetic effect of the lens post insertion, then remove the lens.

SUMMARY:
The study is designed to test five new soft contact lens color pattern variants to determine whether the test lens makes the wearers eyes look bigger, more defined or enhances their overall appearance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age and no more than 39 years of age (inclusive)
2. Subjects must be Asian female
3. Subjects must be able to read Chinese
4. Subjects' monthly household income must be above HKD$ 10,000
5. Subjects must be habitual soft contact lens wearer or habitual limbal lens wearer or have a history of previous habitual lens wear.
6. Subjects' current/previous habitual lens must be in the disposable soft lens modality (ranging from daily to monthly)
7. Subjects must have dark colored iris (black, brown, or brown hazel)
8. Subjects must be "concept acceptors". Concept acceptors are subjects that are willing to try new circle contact lenses.
9. Subjects must be classified as either 'Classic' or 'Vogue' on a Pattern Evaluation Screening Questionnaire.
10. Subjects must have acceptable near vision (without vision correction) and be able to see the test article lenses in the mirror 30 cm or closer.
11. Subjects must have best corrected visual acuity of 20/40 (Snellen or equivalent) or better in each eye.
12. Subjects must possess a functional/usable pair of spectacles and bring them to the visit (only if applicable-to the investigators discretion)
13. Subjects must read, understand, and sign the Statement of Informed Consent
14. Subjects must appear able and willing to adhere to the instructions set forth in this clinical protocol

Exclusion Criteria:

1. Subjects, or subjects' family member within the same household, that work for the following entities/companies: Government, advertising, marketing research or consultancy, media or public relations, companies that make, distribute or sell eyewear or contact lenses, eyecare practice (optometrist, ophthalmologist, optician) or the research center conducting the study
2. Habitual wearers of rigid gas permeable lenses within the last 3 months
3. Habitual soft conventional contact lens wearers (conventional lenses defined as replacement modality of greater than 1 month)
4. Any color deficiencies, by self report
5. Currently pregnant or breast-feeding a baby
6. Diabetes
7. Any ocular or systemic allergies or diseases which may interfere with contact lens wear
8. Any systemic disease, autoimmune disease, or use of medication which may interfere with contact lens wear, at the investigator's discretion
9. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self report
10. Any grade 3 or greater Biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale
11. Any active ocular abnormalities/conditions that may interfere with contact lens wear (this includes, but not limited to, chalazia, recurrent styes, pterygium, infection, etc.)
12. Any corneal distortion or moderate or above corneal distortion by self report
13. History of any corneal refractive surgery
14. Habitual contact lens is multifocal, monovision or worn as extended wear

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Hom, Kowloon, Hong Kong

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 257 subjects were enrolled into this study. Of the enrolled subjects, 240 subjects were dispensed at least 1 study lenses, while 17 subjects failed to meet the eligibility criteria. No subjects were discontinued during the course of this study.
Groups:
- AP-CS-LA-JG-VC; AP-JG-CS-VC-LA; AP-LA-VC-CS-JG; AP-VC-JG-LA-CS; CS-AP-VC-JG-LA; CS-JG-AP-LA-VC; CS-VC-LA-AP-JG; CS-LA-JG-VC-AP; JG-AP-LA-VC-CS; JG-CS-VC-LA-AP; JG-LA-CS-AP-VC; JG-VC-AP-CS-LA; LA-AP-JG-CS-VC; LA-CS-AP-VC-JG; LA-JG-VC-AP-CS; LA-VC-CS-JG-AP; VC-AP-CS-LA-JG; VC-CS-JG-AP-LA; VC-JG-LA-CS-AP; VC-LA-AP-JG-CS: All lenses used in this study were etafilcon A. The lens title correspond to the lens name listed in the protocol registration and refers to various lens variants
Period: Period 1
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least 1 study lens
Groups:
- Total: Total of all reporting groups
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (5.84) | 26.9 (5.78) | 27.9 (4.96) | 28.0 (5.80) | 30.3 (6.06) | 27.5 (4.93) | 28.2 (6.99) | 26.8 (6.58) | 28.9 (5.62) | 26.6 (4.27) | 27.5 (5.04) | 27.3 (5.88) | 29.1 (5.37) | 26.8 (4.37) | 27.85 (5.50) | 26.3 (5.80) | 27.8 (6.29) | 29.9 (6.53) | 27.6 (2.97) | 30.1 (5.11) | 28.0 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 240
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 240
Region of Enrollment [Number; unit: Participants]
  China | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 240

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject in Agreement (Bigger Eyes)
Description: Subjects' responses to the question "Make my eye look bigger" were categorized into a binary variable. If a subject responded "Agrees Somewhat" or "Agrees Strongly" then response=1. If a subject responds "Neither Agrees nor Disagrees", "Disagrees Somewhat" "Disagrees Strongly" then response=0. The number of subjects with response=1 was reported for each lens.
Time Frame: 15-20 Minutes Post Lens Insertion
Population: Subjects that completed all study visits without a major protocol deviation impacting any of the primary endpoints
Measure: Number; unit: Participants
Groups:
- AP- Etafilcon A: Subjects that wore the AP investigational lens during any of the 5 period of the study.
- CS- Etafilcon A: Subjects that wore the CS investigational lens during any of the 5 period of the study.
- JG-etafilcon A: Subjects that wore the JG investigational lens during any of the 5 period of the study.
- LA-etafilcon A: Subjects that wore the LA investigational lens during any of the 5 period of the study.
- VC- Etafilcon A: Subjects that wore the VC investigational lens during any of the 5 period of the study.
Arm/Group | AP- Etafilcon A | CS- Etafilcon A | JG-etafilcon A | LA-etafilcon A | VC- Etafilcon A
Number analyzed (Participants) | 236 | 236 | 236 | 236 | 236
Participants | 187 | 213 | 206 | 209 | 208

2. Primary Outcome: Number of Subject in Agreement (Defines Eyes)
Description: Subjects' responses to the question "Define my eye" were categorized into a binary variable. If a subject responded "Agrees Somewhat" or "Agrees Strongly" then response=1. If a subject responds "Neither Agrees nor Disagrees", "Disagrees Somewhat" "Disagrees Strongly" then response=0. The number of subjects with response=1 was reported for each lens.
Time Frame: 15-20 Minutes Post Lens Insertion
Population: Subjects that completed all study visits without a major protocol deviation impacting any of the primary endpoints
Measure: Number; unit: Participants
Arm/Group | AP- Etafilcon A | CS- Etafilcon A | JG-etafilcon A | LA-etafilcon A | VC- Etafilcon A
Number analyzed (Participants) | 236 | 236 | 236 | 236 | 236
Participants | 175 | 189 | 180 | 188 | 192

3. Primary Outcome: Number of Subject in Agreement (Enhance Eyes)
Description: Subjects' responses to the question "Enhance my overall appearance" were categorized into a binary variable. If a subject responded "Agrees Somewhat" or "Agrees Strongly" then response=1. If a subject responds "Neither Agrees nor Disagrees", "Disagrees Somewhat" "Disagrees Strongly" then response=0. The number of subjects with response=1 was reported for each lens.
Time Frame: 15-20 Minutes Post Lens Insertion
Population: Subjects that completed all study visits without a major protocol deviation impacting any of the primary endpoints
Measure: Number; unit: Participants
Arm/Group | AP- Etafilcon A | CS- Etafilcon A | JG-etafilcon A | LA-etafilcon A | VC- Etafilcon A
Number analyzed (Participants) | 236 | 236 | 236 | 236 | 236
Participants | 167 | 180 | 177 | 170 | 185

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 hours per subject
Arm/Group | AP-CS-LA-JG-VC | AP-JG-CS-VC-LA | AP-LA-VC-CS-JG | AP-VC-JG-LA-CS | CS-AP-VC-JG-LA | CS-JG-AP-LA-VC | CS-VC-LA-AP-JG | CS-LA-JG-VC-AP | JG-AP-LA-VC-CS | JG-CS-VC-LA-AP | JG-LA-CS-AP-VC | JG-VC-AP-CS-LA | LA-AP-JG-CS-VC | LA-CS-AP-VC-JG | LA-JG-VC-AP-CS | LA-VC-CS-JG-AP | VC-AP-CS-LA-JG | VC-CS-JG-AP-LA | VC-JG-LA-CS-AP | VC-LA-AP-JG-CS
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days